CLINICAL TRIAL: NCT07382089
Title: Effect of Oral Hygiene Care on Aspiration Pneumonia Among Hospitalized Stroke Patients: A Quasi-Experimental Study With Historical Controls
Brief Title: Effect of Oral Hygiene Care on Prevention of Aspiration Pneumonia Among Hospitalized Stroke Patients
Acronym: OH-STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Surafel Tilahun Maru, Investigator, Addis Ababa University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASH_OH_STROKE_AP1
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Aspiration Pneumonia
Keywords: Oral hygiene; Aspiration pneumonia prevention; Stroke patients; Dysphagia; Hospital-acquired pneumonia
MeSH Terms: conditions — Stroke; Pneumonia, Aspiration; Deglutition Disorders; Healthcare-Associated Pneumonia | interventions — Oral Hygiene

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, parallel assignment study using historical controls. Patients admitted after implementation of the oral hygiene care protocol received the intervention, while patients admitted prior to implementation served as the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Hygiene Care Intervention (Experimental): Patients admitted after implementation of a structured oral hygiene care protocol delivered by trained nursing staff during hospitalization.
  Interventions: Behavioral: Oral hygiene care bundle
- Historical Control Group (No Intervention): Patients admitted prior to implementation of the oral hygiene care protocol who received standard oral care.

INTERVENTIONS:
Behavioral: Oral hygiene care bundle — A structured oral hygiene care protocol including regular oral cavity cleaning and toothbrushing during hospitalization.
  Other Names: Oral hygiene
  Arms: Oral Hygiene Care Intervention

SUMMARY:
Aspiration pneumonia is a common and serious complication among hospitalized patients with stroke. Poor oral hygiene can increase the risk of aspiration pneumonia by promoting bacterial colonization of the oral cavity. This study evaluated whether implementing a structured oral hygiene care protocol during hospitalization could reduce the incidence of aspiration pneumonia among stroke patients. In this non-randomized, quasi-experimental study, patients admitted after implementation of an oral hygiene care protocol received structured oral care delivered by trained nursing staff, while patients admitted prior to implementation served as historical controls and received standard care. The primary outcome was the occurrence of aspiration pneumonia during hospitalization. The findings of this study aim to inform simple, low-cost preventive strategies that may improve clinical outcomes for hospitalized stroke patients, particularly in resource-limited settings.

DETAILED DESCRIPTION:
This study is a quasi-experimental, non-randomized interventional study with parallel assignment using historical controls, conducted among hospitalized adult stroke patients at a tertiary care hospital. The study evaluated the effect of implementing a structured oral hygiene care protocol on the incidence of aspiration pneumonia during hospitalization. Patients admitted prior to implementation of the oral hygiene care protocol constituted the historical control group and received standard oral care practices. Patients admitted after implementation received a structured oral hygiene care bundle delivered by trained nursing staff as part of routine inpatient care. The oral hygiene intervention included regular oral cavity cleaning and toothbrushing according to a predefined protocol. The primary outcome was aspiration pneumonia diagnosed during hospitalization based on clinical features and radiologic findings. Secondary outcomes included in-hospital clinical outcomes as defined in the study protocol. Ethical approval was obtained from the Institutional Review Board of Tikur Anbessa Specialized Hospital, and informed consent was obtained from participants or their legal representatives, with appropriate waivers applied for retrospective data where applicable. This study was designed to assess the feasibility and effectiveness of a low-cost, preventive intervention that may reduce aspiration-related complications among stroke patients, particularly in resource-constrained healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Hospitalized patients with a confirmed diagnosis of acute stroke (ischemic or hemorrhagic)
* Admission to the stroke unit or medical ward during the study period
* Ability to receive oral care as part of routine nursing care

Exclusion Criteria:

* Patients with active pneumonia at the time of hospital admission
* Patients who were intubated or mechanically ventilated at admission
* Patients with facial or oral conditions precluding oral hygiene care
* Patients discharged or deceased within 24 hours of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Aspiration Pneumonia | From baseline (hospital admission) through hospital discharge, up to 21 days
  Aspiration pneumonia diagnosed during hospital admission, based on clinical features (fever, cough, purulent sputum), radiologic evidence of new pulmonary infiltrates, and treating physician documentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tikur Anbessa Specialized Hospital, Addis Ababa University, Addis Ababa, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen HJ, Chen JL, Chen CY, Lee M, Chang WH, Huang TT. Effect of an Oral Health Programme on Oral Health, Oral Intake, and Nutrition in Patients with Stroke and Dysphagia in Taiwan: A Randomised Controlled Trial. Int J Environ Res Public Health. 2019 Jun 24;16(12):2228. doi: 10.3390/ijerph16122228. PMID 31238591
- [Result] O'Malley L, Powell R, Hulme S, Lievesley M, Westoby W, Zadik J, Bowen A, Brocklehurst P, Smith CJ. A qualitative exploration of oral health care among stroke survivors living in the community. Health Expect. 2020 Oct;23(5):1086-1095. doi: 10.1111/hex.13074. Epub 2020 Jun 19. PMID 32558061
- [Result] Dai R, Lam OLT, Lo ECM, Li LSW, McGrath C. A randomized clinical trial of oral hygiene care programmes during stroke rehabilitation. J Dent. 2017 Jun;61:48-54. doi: 10.1016/j.jdent.2017.04.001. Epub 2017 Apr 6. PMID 28392215
- [Result] Kim EK, Park EY, Sa Gong JW, Jang SH, Choi YH, Lee HK. Lasting effect of an oral hygiene care program for patients with stroke during in-hospital rehabilitation: a randomized single-center clinical trial. Disabil Rehabil. 2017 Nov;39(22):2324-2329. doi: 10.1080/09638288.2016.1226970. Epub 2016 Sep 15. PMID 27628624
- [Result] Chan EY, Lee YK, Poh TH, Ng IH, Prabhakaran L. Translating evidence into nursing practice: oral hygiene for care dependent adults. Int J Evid Based Healthc. 2011 Jun;9(2):172-83. doi: 10.1111/j.1744-1609.2011.00214.x. PMID 21599846
- [Result] Cardoso AF, Ribeiro LE, Santos T, Pinto M, Rocha C, Magalhaes J, Augusto B, Santos D, Duque FM, Fernandes BL, Sousa RC, Silva R, Ventura F, Fernandes AM, Cardoso D, Rodrigues R. Oral Hygiene in Patients with Stroke: A Best Practice Implementation Project Protocol. Nurs Rep. 2023 Jan 31;13(1):148-156. doi: 10.3390/nursrep13010016. PMID 36810267